CLINICAL TRIAL: NCT06885593
Title: "Can Femoral Vena Cava Collapsibility Index Predict Post-spinal Hypotension in Pregnant Women in Left Lateral Tilt Position?"
Brief Title: Femoral Vein Collapsibility Index and Post-Spinal Hypotension in Pregnant Women: Impact of Position
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mehmet Sarı (Other)
Responsible Party: Sponsor-Investigator, Mehmet Sarı, Principal Investigator, Bezmialem Vakif University
Organization: Bezmialem Vakif University (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2025/7
Record Dates: First submitted 2025-03-10; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Spinal Induced Hypotension in Cesarean Delivery
MeSH Terms: interventions — Supine Position

STUDY DESIGN:
Intervention Model Description: All ultrasonography (USG) procedures will be performed by the same anesthesiologist using a Ultrasound device before the start of spinal anesthesia (SA) and after baseline blood pressure and heart rate have been measured. Patients will be placed in supine and left lateral tilt (LLT) positions. After at least 3 minutes in each position, ultrasound of the inferior vena cava (IVC) and femoral vein (FV) will be performed. The oblique probe will be placed below the xiphoid. Anteroposterior diameters and peak velocities of the IVC will be measured 2-3 cm below the IVC-right atrium For standardization purposes, measurements of the right femoral vein will be used in the study. The FV will be visualized with B-mode ultrasound 2-5 cm below the level of the inguinal ligament where the femoral artery is best palpated, without applying any pressure that may affect the FV diameter.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: In this clinical trial, besides the anesthesiologist performing the ultrasonography (USG), the following parties will be masked:
  Outcome Assessor(s): The individuals responsible for measuring the post-spinal hypotension outcomes, such as blood pressure and heart rate, will be blinded to the patient's assigned position (supine or left lateral tilt). This ensures that their measurements and assessments are not influenced by the positioning during the ultrasound evaluation.
  Data Analysts: The data analysts, who will perform the statistical analysis of the study outcomes, will be blinded to the group assignments (supine or left lateral tilt). This is done to avoid bias in interpreting the results related to the position and its effect on post-spinal hypotension.
  Patients: The patients themselves will not be aware of the specific position (supine or left lateral tilt) they are assigned to during the ultrasound procedure, as this will be randomized. However, they will be informed of the pro
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Supine Position (Sham Comparator): All ultrasonography (USG) procedures will be performed by the same anesthesiologist using a Ultrasound device before the start of spinal anesthesia (SA) and after baseline blood pressure and heart rate have been measured. Patients will be placed in supine position. After at least 3 minutes in each position, ultrasound of the inferior vena cava (IVC) and femoral vein (FV) will be performed. The oblique probe will be placed below the xiphoid. Anteroposterior diameters and peak velocities of the IVC will be measured 2-3 cm below the IVC-right atrium For standardization purposes, measurements of the right femoral vein will be used in the study. The FV will be visualized with B-mode ultrasound 2-5 cm below the level of the inguinal ligament where the femoral artery is best palpated, without applying any pressure that may affect the FV diameter.
  Interventions: Diagnostic Test: Supine Position; Diagnostic Test: Left Lateral Tilt Position
- Left Lateral Tilt Position (Active Comparator): All ultrasonography (USG) procedures will be performed by the same anesthesiologist using a Ultrasound device before the start of spinal anesthesia (SA) and after baseline blood pressure and heart rate have been measured.
  Patients will be placed in left lateral tilt (LLT) positions. After at least 3 minutes in each position, ultrasound of the inferior vena cava (IVC) and femoral vein (FV) will be performed. The oblique probe will be placed below the xiphoid. Anteroposterior diameters and peak velocities of the IVC will be measured 2-3 cm below the IVC-right atrium For standardization purposes, measurements of the right femoral vein will be used in the study. The FV will be visualized with B-mode ultrasound 2-5 cm below the level of the inguinal ligament where the femoral artery is best palpated, without applying any pressure that may affect the FV diameter.
  Interventions: Diagnostic Test: Supine Position; Diagnostic Test: Left Lateral Tilt Position

INTERVENTIONS:
Diagnostic Test: Supine Position — All ultrasonography (USG) procedures will be performed by the same anesthesiologist using a Ultrasound device before the start of spinal anesthesia (SA) and after baseline blood pressure and heart rate have been measured. Patients will be placed in supine and left lateral tilt (LLT) positions. After at least 3 minutes in each position, ultrasound of the inferior vena cava (IVC) and femoral vein (FV) will be performed. The oblique probe will be placed below the xiphoid. Anteroposterior diameters and peak velocities of the IVC will be measured 2-3 cm below the IVC-right atrium For standardization purposes, measurements of the right femoral vein will be used in the study. The FV will be visualized with B-mode ultrasound 2-5 cm below the level of the inguinal ligament where the femoral artery is best palpated, without applying any pressure that may affect the FV diameter.
Diagnostic Test: Supine Position — All ultrasonography (USG) procedures will be performed by the same anesthesiologist using a Ultrasound device before the start of spinal anesthesia (SA) and after baseline blood pressure and heart rate have been measured. Patients will be placed in supine position. After at least 3 minutes in each position, ultrasound of the inferior vena cava (IVC) and femoral vein (FV) will be performed. The oblique probe will be placed below the xiphoid. Anteroposterior diameters and peak velocities of the IVC will be measured 2-3 cm below the IVC-right atrium For standardization purposes, measurements of the right femoral vein will be used in the study. The FV will be visualized with B-mode ultrasound 2-5 cm below the level of the inguinal ligament where the femoral artery is best palpated, without applying any pressure that may affect the FV diameter.
Diagnostic Test: Left Lateral Tilt Position — All ultrasonography (USG) procedures will be performed by the same anesthesiologist using a Ultrasound device before the start of spinal anesthesia (SA) and after baseline blood pressure and heart rate have been measured. Patients will be placed in left lateral tilt (LLT) position. After at least 3 minutes in each position, ultrasound of the inferior vena cava (IVC) and femoral vein (FV) will be performed. The oblique probe will be placed below the xiphoid. Anteroposterior diameters and peak velocities of the IVC will be measured 2-3 cm below the IVC-right atrium For standardization purposes, measurements of the right femoral vein will be used in the study. The FV will be visualized with B-mode ultrasound 2-5 cm below the level of the inguinal ligament where the femoral artery is best palpated, without applying any pressure that may affect the FV diameter.

SUMMARY:
This study aims to improve the safety of spinal anesthesia for pregnant patients undergoing elective cesarean delivery. Specifically, the investigators are investigating whether ultrasound measurements of a vein in the groin (the right common femoral vein, or RCFV) can help predict the risk of low blood pressure (hypotension) after spinal anesthesia. The main question it aims to answer is:

Can femoral vena cava collapsibility index predict post-spinal hypotension in pregnant women in left lateral tilt position?

Before receiving spinal anesthesia, participants will undergo a brief and painless ultrasound examination of the RCFV in the groin area while lying in a specific position."

DETAILED DESCRIPTION:
Post-spinal hypotension (PSH) is defined as a systolic arterial blood pressure (SBP) decrease of more than 20% from baseline or an SBP drop below 100 mmHg. This reduction in blood pressure may compromise uteroplacental perfusion, leading to fetal hypoxia and acidosis. PSH is the most common complication in obstetric anesthesia, with an incidence of up to 95% in healthy women. Despite extensive research, the most effective strategy to maintain hemodynamic stability remains under investigation. Various methods, including crystalloid and colloid fluid loading, leg wrapping, head-down tilt, and vasopressor use, have been explored for both treatment and prevention.

The sympatholytic effect of spinal anesthesia induces vasodilation, exacerbating maternal hypotension due to the gravid uterus compressing the inferior vena cava (IVC). This compression reduces venous return and subsequently decreases the IVC diameter.

Current recommendations for term pregnant women undergoing cesarean delivery advocate for a left lateral tilt position to prevent aortocaval compression (ACC), maternal hypotension, and fetal compromise . In the supine position, the IVC is nearly completely obstructed at term up to its bifurcation. However, most women experience only minimal hemodynamic effects due to compensatory mechanisms such as venoconstriction in the lower extremities and collateral circulation via the paraspinal and azygos veins. Clinically significant hemodynamic compromise, known as supine hypotensive syndrome, occurs in approximately 8-10% of term pregnancies, likely due to insufficient compensatory responses .

The right common femoral vein (RCFV), a continuation of the right external iliac vein, is a tributary of the IVC. Because the RCFV is superficially located, it can be easily visualized using a high-frequency ultrasound probe. Importantly, the RCFV is situated distal to the site of aortocaval compression, making it a potential surrogate marker for hemodynamic changes.

Study Hypothesis This study hypothesizes that the peak velocity and collapsibility index of the RCFV in the inguinal region, measured in the left lateral 15-degree tilt position, reflect the degree of aortocaval compression. These parameters may help identify pregnant women at high risk of post-spinal hypotension during elective cesarean delivery.

ELIGIBILITY:
Inclusion Criteria:

* ASA 2
* Uncomplicated pregnancy
* Height between 150 cm-180 cm
* Signed the informed consent form
* 8 hours of fasting before the operation
* Patients who refuse normal delivery

Exclusion Criteria:

* Obstetric comorbidities affecting caval compression of the aorta
* Transverse development
* Fetal macrosomia
* Uterine anomaly
* Polyhydramnion
* Oligohydroamnion
* Membrane ruptures
* Intrauterine growth retardation
* Mothers with hyperactive lung disease
* Those with autonomic neuropathy
* Kidney failure
* Smokers
* Severe scoliosis or kyphosis
* Multiple pregnancy (twins, triplets,...)
* Those who do not reach T6 sensory block level after 10 minutes
* Those undergoing general anesthesia or IV analgesics for any reason

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Post-Spinal Hypotension | 40 minute
  Post-Spinal Hypotension Measured by Systolic and Diastolic Blood Pressure and Heart Rate Changes Following Spinal Anesthesia in Supine and Left Lateral Tilt Positions Systolic Blood Pressure, Diastolic Blood Pressure, and Heart Rate are now presented as separate outcome measures, each with its own unit of measure.

SECONDARY OUTCOMES:
Number of Participants with time of onset of maternal hypotension, symptomatic hypotension, incidence of bradycardia, cumulative ephedrine requirements, patient satisfaction | 24 hours
  Secondary maternal outcomes recorded from the induction of spinal anesthesia (SA) to delivery include: time of onset of maternal hypotension (time from SA to first hypotension episode); symptomatic hypotension (hypotension with nausea, vomiting, and/or dizziness); severe hypotension (systolic arterial pressure [SAP] <70% of baseline); minimum recorded SAP; cumulative duration of hypotension (total minutes of SAP <90 mmHg or diastolic BP <60 mmHg); minimum heart rate (HR); incidence of bradycardia (HR <50 bpm); atropine use for bradycardia; cumulative ephedrine requirements (total ephedrine dose administered); and patient satisfaction (rated on a Likert scale from 1-5).

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakıf Univeristesi Dragos Hastanesi Yalı, Kennedy Cd. No:16., Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yao SF, Zhao YH, Zheng J, Qian JY, Zhang C, Xu Z, Xu T. The transverse diameter of right common femoral vein by ultrasound in the supine position for predicting post-spinal hypotension during cesarean delivery. BMC Anesthesiol. 2021 Jan 20;21(1):22. doi: 10.1186/s12871-021-01242-8. PMID 33472587
- [Background] Lal J, Jain M, Rahul, Singh AK, Bansal T, Vashisth S. Efficacy of inferior vena cava collapsibility index and caval aorta index in predicting the incidence of hypotension after spinal anaesthesia- A prospective, blinded, observational study. Indian J Anaesth. 2023 Jun;67(6):523-529. doi: 10.4103/ija.ija_890_22. Epub 2023 Jun 14. PMID 37476444